CLINICAL TRIAL: NCT00060112
Title: A Phase I Study of Oblimersen (Genasense™, G3139) in Combination With Gemcitabine in Advanced Malignancies
Brief Title: Oblimersen and Gemcitabine in Treating Patients With Advanced Solid Tumor or Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02531; SUMC-78808; CDR0000299507 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Splenic Marginal Zone Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — oblimersen; Gemcitabine

ARMS (1):
- Treatment (oblimersen sodium and gemcitabine hydrochloride) (Experimental): Patients receive oblimersen IV continuously on days 1-5 and gemcitabine IV over 2-3 hours on day 5. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: oblimersen sodium; Drug: gemcitabine hydrochloride; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: oblimersen sodium — Given IV
  Other Names: augmerosen; G3139; G3139 bcl-2 antisense oligodeoxynucleotide; Genasense
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy such as gemcitabine use different ways to stop cancer cells from dividing so they stop growing or die. Oblimersen may increase the effectiveness of gemcitabine by making cancer cells more sensitive to the drug. This phase I trial is studying the side effects and best dose of oblimersen and gemcitabine in treating patients with metastatic or unresectable solid tumors or lymphoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose and dose-limiting toxicity of oblimersen and gemcitabine in patients with advanced solid tumor or lymphoma.

II. Determine the effect of oblimersen on the pharmacokinetics and pharmacodynamics of gemcitabine in these patients.

III. Determine the toxic effects of this regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive oblimersen IV continuously on days 1-5 and gemcitabine IV over 2-3 hours on day 5. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of oblimersen and gemcitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Up to 10 additional patients receive treatment at the MTD.

PROJECTED ACCRUAL: Approximately 15 patients will be accrued for this study within 6-8 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy for which there is no standard or effective curative or palliative therapy

  * Solid tumors and lymphoma allowed
  * Metastatic or unresectable disease
* Measurable or evaluable nonmeasurable disease

  * Evaluable nonmeasurable disease includes ascites, pleural/pericardial effusions, lymphangitis cutis/pulmonis, inflammatory breast disease, abdominal masses not followed by CT scan or MRI, or cystic lesions
  * Disease characterized by elevated serum tumor marker alone is allowed
* No known brain metastases
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 3 months
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 mg/dL
* AST and ALT no greater than 2.5 times upper limit of normal
* No history of portal hypertension
* No history of cirrhosis or hepatitis
* No radiographic evidence of cirrhosis and/or varices
* Creatinine normal
* Creatinine clearance at least 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to oblimersen or other study agents
* No other concurrent uncontrolled illness that would preclude study participation
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No concurrent prophylactic colony-stimulating factors such as filgrastim (G-CSF) or sargramostim (GM-CSF)
* Concurrent interventional growth factors allowed

  * No growth factor administration within 24 hours before study chemotherapy
* Concurrent epoetin alfa allowed
* No more than 3 prior chemotherapy regimens
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* More than 2 weeks since prior hormonal therapy
* Concurrent megestrol for anorexia/cachexia allowed
* No prior pelvic or whole abdominal radiotherapy
* More than 4 weeks since prior radiotherapy
* More than 4 weeks since prior major surgery
* Recovered from prior therapy
* More than 4 weeks since prior investigational therapy
* No prior oblimersen
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-03; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose level at which less than 2 out of 6 patients experience DLT assessed using NCI CTC version 2.0 | 4 weeks
  Descriptive statistics will be employed in the analysis of all safety and laboratory observations.

SECONDARY OUTCOMES:
Pharmacokinetics | Pre-dose, 4, 8, 12, 24, 48, 72, 96, 120, 121.67, 126, and 129 hours
  Peak concentration and area under the concentration time curves of gemcitabine triphosphate will be will be utilized to assess the pharmacodynamic relationship of gemcitabine triphosphate concentration to bivariate toxicity and tumor responses using logistic regression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Branimir (Brandy) Sikic, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States